CLINICAL TRIAL: NCT00855998
Title: Thymidine Kinase 1 in Risk Assessment for Hereditary Breast /Ovarian Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Prof. Tamar Peretz, Head of Oncology Department, Hadassah Medical Organization
Other Study IDs: 044608-HMO-CTIL
Record Dates: First submitted 2009-02-22; First posted 2009-03-05 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2009-03

CONDITIONS: Breast Cancer; Ovarian Cancer
Keywords: Thymidine Kinase 1; BRCA1 and BRCA2 mutations; hereditary breast/ovarian cancer
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: With BRCA1 or BRCA2 mutations
- 2: Without BRCA1 or BRCA2 mutations

SUMMARY:
This study aimed to compare the activity of Thymidine Kinase 1 in serum of two groups of woman at high and normal risk for breast/ovary cancer.

DETAILED DESCRIPTION:
Hereditary breast/ovarian cancer syndrome is associated with mutations in tumor suppressor BRCA1 and BRCA2 genes. Products of these genes play an important role in the repair of DNA double-strand breaks. Mutations in BRCA1 and BRCA2 genes could impair DNA repair. In resting or G1 cells, where the de novo synthesis of DNA precursors is absent, the salvage pathway is the sole provider of deoxyribonucleotides to be used in DNA repair. For this process a sufficient supply of deoxynucleotides and activity of Thymidine Kinase 1 are essential. TK1 is an important component of adaptive response of cells to DNA damage. Mutations in genes directly engaged in the DNA repair process could lead to the accumulation of DNA damage and in turn cause an adaptive cell reaction manifesting as permanently increased Thymidine Kinase 1 activity.

A recently developed new high-sensitive assay DiviTum® allows to investigate the contribution of this enzyme to DNA repair processes and to make a comparison of Thymidine kinase 1 activity in women with normal and impared DNA repair system.

ELIGIBILITY:
Inclusion Criteria:

* women from family with more than two breast cancer cases and one or more cases of ovarian cancer diagnosed at any age;
* women from family with more than three breast cancer cases diagnosed before the age 50;
* women from family withsister pair in which one of the following combinations was diagnosed before the age of 50: two breast cancers, two ovarian cancers, or a breast and ovarian cancer.

Exclusion Criteria:•

* pregnant women;
* women with generalized CMV and HZV infections;
* women with severe B12 deficiency and megaloblastic anaemia;
* women with severe rheumatoid arthritis.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: women visiting the outpatient oncology clinic for genetic/familial high-risk assessments
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-03 (Estimated); Study Completion 2011-03 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Derived] Nisman B, Kadouri L, Allweis T, Maly B, Hamburger T, Gronowitz S, Peretz T. Increased proliferative background in healthy women with BRCA1/2 haploinsufficiency is associated with high risk for breast cancer. Cancer Epidemiol Biomarkers Prev. 2013 Nov;22(11):2110-5. doi: 10.1158/1055-9965.EPI-13-0193. Epub 2013 Aug 21. PMID 23966579